CLINICAL TRIAL: NCT05261529
Title: Effects of a Nutricional Intervention With EVOO Oil and Physical Activity in Patients With Systemic Lupus Erythematosus: Effect on Clinical Course, Epigenetic and Microbiome
Brief Title: Effects of an Intervention With EVOO and Physical Activity in Patients With Systemic Lupus Erythematosus
Acronym: EFINUTRILES
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad de Granada (Other)
Collaborators: Consejería de Economía, Innovación y Ciencia. Proyectos de I+D+I en el marco operativo Feder Andalucía 2014-2020 (Unknown)
Responsible Party: Principal Investigator, María Correa-Rodríguez, Associate Professor, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2099-N-21
Record Dates: First submitted 2022-02-08; First posted 2022-03-02 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Lupus Erythematosus, Systemic
Keywords: Mediterranean Diet; Olive Oil; Physical Exercise; Autoimmune Diseases; Systemic Lupus Erythematosus; Microbiome; Epigenetcis
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Motor Activity; Autoimmune Diseases

STUDY DESIGN:
Intervention Model Description: Three-arm prospective randomized controlled 24-week clinical trial of patients diagnosed with SLE.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Participants randomly assigned in a 1:1:1 ratio to each of the three groups established through a centralized method with computer support (OxMaR software).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (No Intervention): Control Group with 30 patients diagnosed with SLE following their normal lifestyle in terms of dietary intake and physical exercise.
- Oil Group (Experimental): Group with 30 patients diagnosed with SLE that add to their normal dietary intake a supplementation with 40ml of EVOO daily during 24 weeks, without changing their lifestyle in terms of physical exercise.
  Interventions: Dietary Supplement: Extra Virgin Olive Oil (EVOO)
- Oil + Exercise Group (Experimental): Group with 30 patients diagnosed with SLE that besides adding to their normal dietary intake a supplementation with 40ml of EVOO daily during 24 weeks, will follow a physical exercise multimodal program the 12 last weeks.
  Interventions: Dietary Supplement: Extra Virgin Olive Oil (EVOO); Behavioral: Physical Exercise Program

INTERVENTIONS:
Dietary Supplement: Extra Virgin Olive Oil (EVOO) — Daily intake of 40ml EVOO added to the normal intake of EVOO of the participants.
  Arms: Oil + Exercise Group; Oil Group
Behavioral: Physical Exercise Program — Besides the EVOO supplementation in the same conditions as the 'Intervention 1 Group', participants will add the follow-up of a Multimodal Physical Exercise (MFE) program during the remaining 12 weeks of intervention, 3 days per week, online and face-to-face group sessions on non-consecutive days. Continuous and intervalic cardiovascular exercise at moderate-intense intensity, controlled by the HR in reserve, with a duration of 15-45 minutes, also including sympathetic modulation exercises (stretching, breathing and meditation) and methods to promote recovery, with a duration of 10-30 minutes.
  Arms: Oil + Exercise Group

SUMMARY:
In addition to the different pharmacological therapies available for the treatment of Systemic Lupus Erythematosus (SLE) as well as for its numerous associated complications (cutaneous, articular, hematological, neuropsychiatric, renal...), it has recently been proposed that 'health-related lifestyles' could have a determining role in balancing numerous organic processes at all levels. In line with this, the benefits of following a healthy dietary pattern such as the Mediterranean Diet and, specifically, the intake of Extra Virgin Olive Oil (EVOO) as well as the realization of regular physical exercise (PE) have been examined in numerous chronic non-communicable diseases such as obesity or cancer. However, in patients with autoimmune diseases, such as SLE, the possible effects of this synergy has not been investigated to date. Having demonstrated both the protective effect of a healthy dietary pattern and that of regular PE on the progression and risks associated with SLE in cross-sectional studies, non-intervention research has been developed that combines both strategies simultaneously, with nutritional supplementation or PE occurring independently. It is hypothesized that supplementation with EVOO in these patients together with PE will produce superior benefits compared to EVOO supplementation alone, showing changes in the phenotype of SLE and other parameters such as levels of chronicity/gravity, biomarkers (oxidative stress, immunological, inflammation), cardiovascular status and body composition.

DETAILED DESCRIPTION:
SLE is one of the more representative autoimmune diseases that courses with several manifestations which are cutaneous-mucosal, joint, hematologic, neuropsychiatric and/or renal. In addition to the different pharmacological therapies available for its treatment, the adequate management of 'health-related lifestyles' becomes a relevant strategy by balancing, among others, the dysbiosis of the microbiota, the production of metabolites and the alteration of the immune response, with positive repercussions on all organic processes. Mediterranean Diet (MD), and the intake of EVOO in specific, which is its most representative food, has been shown to be a proven dietary pattern of protection against chronic non-communicable diseases. In line with this, Physical Exercise (PE) is another strategy on the rise. Regular exercise at moderate intensity has great impact on the immune system, the central nervous system, as a regulator of hormones and blood glucose levels, and on the psychosocial and cognitive spheres, ultimately leading to the appearance of numerous beneficial modifications in the face of external pathogenic aggressions and inflammatory processes.

Therefore, the synergy between DM and PE could enhance the known beneficial effects of both types of approaches in patients with SLE, as the scientific literature has shown in other chronic diseases such as obesity or cancer, among others. However, there are currently few studies that include PE interventions, and there is also some contradiction in the results. In addition, there is no study that synergizes both approaches in a coincident manner over time. The present study, whose main objective is to analyze the influence of the addition to a supplementation with EVOO of a multimodal combined physical exercise intervention in patients with SLE, is developed under the hypothesis that: The combination of dietary supplementation with EVOO together with the follow-up of a multimodal PE program will result in superior benefits in SLE patients with respect to a group of patients solely supplemented with EVOO, showing changes in SLE phenotype and parameters such as levels of chronicity/severity of the disease, levels of biochemical, immunological, inflammatory and oxidative stress markers, markers of cardiovascular risk and early atherosclerosis and endothelial function, cardiorespiratory status and body composition.

For this purpose, a 24-week clinical trial will be developed with three groups of patients with SLE (30 patients/group): a control group (no intervention), another that will add to the usual intake pattern of 40ml of EVOO daily during 24 weeks, and a third group that will add to this additional intake of EVOO the follow-up of a specific PE program in the middle of the intervention (12 weeks).

Data collection in all groups will be perform before the intervention, at an intermediate stage and coinciding with the beginning of the PE program (12 weeks), and at the end of the study (24 weeks).

The study will be carried out in three phases:

STAGE 1: Reinforcement of adherence to DM. In order to guarantee during the intervention the maintenance of the levels of adherence to DM established as inclusion criteria, previously and in both groups the basic principles of DM will be recalled by a nutritionist, through group sessions of 1 hour of duration.

STAGE 2: Intervention. EVOO supplementation, or EVOO supplementation + PE under the conditions previously described. The intervention, which will be extended over 24 weeks, will consist of the daily consumption of 40 ml of EVOO in a single daily intake, added to the usual intake pattern of the participants.

* CG. The participants' usual lifestyle (dietary pattern and physical activity) will not be modified.
* Intervention Group 1. Patients will take the EVOO supplementation as describe below, without changing their physical activity routines.
* Intervention Group 2. In addition to taking EVOO supplementation, patients will start following a Multimodal Physical Exercise (MFE) program during the remaining 12 weeks of intervention, guided by personnel with experience in the area: 3 days per week, groupal sessions (≤10 participants/group) on non-consecutive days, both online and face-to-face sessions. Continuous (4-6weeks) and intervallic (week 5-7 to 24) cardiovascular exercise will be worked at moderate-intense intensity, controlled by HR in reserve, with a duration of 15-45 minutes. In addition, sympathetic modulation exercises (stretching, breathing, meditation) will be used as methods to promote recovery, with a duration of 10-30 minutes. In this group, supplementation will take place after exertion.

STAGE 3: Post-intervention data collection (week 25).

ELIGIBILITY:
Patients will be eligible if they have been diagnosed with SLE for at least one year and have been seen at the Outpatient Clinic of the Systemic Autoimmune Diseases Unit of the Hospital Universitario Clínico San Cecilio of Granada (Spain), meet the revised American College of Rheumatology (ACR), SLICC or ACR/EULAR criteria of 2019 and maintain a stable SLEDAI-2K, without treatment modifications, in the previous 3 months.

Inclusion Criteria:

* Medium (8 to 11 points) to high (12 to 14 points) level of adherence to DM as measured by the 14-point DM adherence scale of the PREDIMED study.
* Sedentary, inactive or non-performing subjects of structured PE (+5h sitting or doing less than 300min of weekly physical activity or <60min structured exercise per week).

Exclusion Criteria:

* Terminal stages of the disease
* Serum creatinine levels ≥1.5mg / dl
* Type 1 Diabetes Mellitus
* Infection, trauma or surgery six months prior to intervention
* SLICC> 5
* Pregnant, with intention, or breastfeeding
* Diagnosis of other autoimmune / inflammatory diseases
* Participation in other PE guided programs
* Contraindication for PE: psychiatric or cognitive disorders, acute or chronic conditions (advanced lung disease, high requirements, stenosis> 70%)
* BMI of morbid obesity (≥40)

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-11-03 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
SLEDAI Systemic Lupus Erythematosus Disease Activity Index | Participants will be followed over 24 weeks.
  SLE-specific index that assess disease activity through a combination of data from clinical records, physical examination, organ-specific functional tests and serological studies.

SECONDARY OUTCOMES:
Cumulative manifestations | Participants will be followed over 24 weeks.
  All the manifestations and complications that patients go through or appear during the intervention, recorded by interview with clinicians.
SLICC/ACR (Systemic Lupus International Collaborating clinics/American College of Rheumatology) Damage Index for Systemic Lupus Erythematosus. | Participants will be followed over 24 weeks.
  Index developed to quantify damage that has occurred since onset of lupus, correlates with mortality. Score and clinical relevance registered by interview with clinicians.
Pharmacological prescription | Participants will be followed over 24 weeks.
  All the medicines that the patients are taking, start to take, o stop taking during the intervention, registered by interview with clinicians.
Glucose level | Participants will be followed over 24 weeks.
  Glucose will be analyzed through blood test.
Urea level | Participants will be followed over 24 weeks.
  Urea will be analyzed through blood test.
Creatinine level | Participants will be followed over 24 weeks.
  Creatinine will be analyzed through blood test.
Lipid profile analysis | Participants will be followed over 24 weeks.
  Lipid profile will be analyzed through blood test.
Creatine Kinase concentration | Participants will be followed over 24 weeks.
  Creatine Kinase (CK) will be analyzed through blood test.
Hemoglobin concentration | Participants will be followed over 24 weeks.
  Hemoglobin (Hb) will be analyzed through blood test.
Number of lymphocytes | Participants will be followed over 24 weeks.
  Number of lymphocytes will be analyzed through blood test.
Number of platelets | Participants will be followed over 24 weeks.
  Number of platelets will be analyzed through blood test.
Number of leukocytes | Participants will be followed over 24 weeks.
  Number of leukocytes will be analyzed through blood test.
Inflammation | Participants will be followed over 24 weeks.
  C-Reactive Protein (CRP) will be analyzed trough blood test.
Anti phospholipid antibodies concentration | Participants will be followed over 24 weeks.
  Autoimmunity Anti phospholipid antibodies parameter will be analyzed through blood test.
Double-stranded anti-DNA antibodies concentration | Participants will be followed over 24 weeks.
  Autoimmunity Double-stranded anti-DNA antibodies parameter will be analyzed through blood test.
Complement fraction C3 concentration | Participants will be followed over 24 weeks.
  Autoimmunity Complement fraction C3 parameter will be analyzed through blood test.
Complement fraction C4 concentration | Participants will be followed over 24 weeks.
  Autoimmunity Complement fraction C4 parameter will be analyzed through blood test.
Cardiorespiratory Fitness | Participants will be followed over 24 weeks.
  Evaluated by Treadmill Ergometric test.
Functional capacity | Participants will be followed over 24 weeks.
  Evaluated by the 6-Minute walking test.
Hight | Participants will be followed over 24 weeks.
  In centimeters; will be evaluated using a measuring tape.
Weight | Participants will be followed over 24 weeks.
  In kilograms; will be evaluated using an Inbody.
Skeletal Muscle Mass | Participants will be followed over 24 weeks.
  In kilograms; will be evaluated using an Inbody.
Body Fat Mass | Participants will be followed over 24 weeks.
  In kilograms; will be evaluated using an Inbody.
Body Mass Index | Participants will be followed over 24 weeks.
  Weight and height will be combined to report Body Mass Index (BMI) in kg/m^2
Body Fat Index | Participants will be followed over 24 weeks.
  In %; will be evaluated using an Inbody.
Waist-to-hip ratio in centimeters | Participants will be followed over 24 weeks.
  In centimeters; waist circumference and hip circumference measures will be combined to calculate waist-to-hip ratio (WHR).
Obesity degree | Participants will be followed over 24 weeks.
  In %; will be evaluated using an Inbody.
Body Cell Mass | Participants will be followed over 24 weeks.
  In kilograms; will be evaluated using an Inbody.
Bone Mineral Content | Participants will be followed over 24 weeks.
  In kilograms; will be evaluated using an Inbody.
Basal Metabolic Rate | Participants will be followed over 24 weeks.
  In kilocalories; will be evaluated using an Inbody.
Visceral Fat Area | Participants will be followed over 24 weeks.
  In cm^2; Visceral Fat Area (AVG) will be evaluated using an Inbody.
Bone density | Participants will be followed over 24 weeks.
  Evaluated by densitometry.
Human Vascular Cell Adhesion Molecule-1 concentration | Participants will be followed over 24 weeks.
  VCAM-1 endothelial biomarker will be assessed by blood test.
Intercellular Adhesion Molecule-1concentration | Participants will be followed over 24 weeks.
  ICAM-1 endothelial biomarker will be assessed by blood test.
E-Selectin concentration | Participants will be followed over 24 weeks.
  E-Selectin endothelial biomarker will be assessed by blood test.
Super Oxide Dismutase concentration | Participants will be followed over 24 weeks.
  Oxidative Stress SOD biomarker will be assessed by blood test.
Glutathione concentration | Participants will be followed over 24 weeks.
  Oxidative Stress GSH biomarker will be assessed by blood test.
Total Antioxidant Capacity concentration | Participants will be followed over 24 weeks.
  Oxidative Stress TAC biomarker will be assessed by blood test.
Thiobarbituric Acid Reactive Substances concentration | Participants will be followed over 24 weeks.
  Oxidative Stress TBARS biomarker will be assessed by blood test.
Malondialdehyde concentration | Participants will be followed over 24 weeks.
  Oxidative Stress MDA biomarker will be assessed by blood test.
Advanced Oxidation Protein Products concentration | Participants will be followed over 24 weeks.
  Oxidative Stress AOPP biomarker will be assessed by blood test.
Total proteins concentration | Participants will be followed over 24 weeks.
  Oxidative Stress total proteins biomarker, understood as the concentration of proteins in a sample, will be assessed by blood test.
Endothelial Function | Participants will be followed over 24 weeks.
  Several endothelial function parameters such are arterial pulse wave velocity, AIX index, ABI will be evaluated using arteriography.
miRNA expression profile quantification | Participants will be followed over 24 weeks.
  Collection of blood samples in Tempus tubes for subsequent analysis of miRNA expression profile by massive sequencing with specific equipment.
Microbiome characteristics analysis | Participants will be followed over 24 weeks.
  Microbiome study by collecting fecal samples.

CONTACTS AND LOCATIONS:
Overall Officials: María Correa Rodríguez, Professor, Principal Investigator — Universidad de Granada
Locations (1):
- Universidad de Granada, Granada, Granada, Spain, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pocovi-Gerardino G, Correa-Rodriguez M, Callejas-Rubio JL, Rios-Fernandez R, Martin-Amada M, Cruz-Caparros MG, Rueda-Medina B, Ortego-Centeno N. Beneficial effect of Mediterranean diet on disease activity and cardiovascular risk in systemic lupus erythematosus patients: a cross-sectional study. Rheumatology (Oxford). 2021 Jan 5;60(1):160-169. doi: 10.1093/rheumatology/keaa210. PMID 32594173
- [Derived] Gil-Gutierrez R, Medina-Martinez I, Quesada-Caballero M, de la Hera-Fernandez FJ, Zamora-Pasadas M, Cantarero-Villanueva I, Albendin-Garcia L, Parola V, Rueda-Medina B, Correa-Rodriguez M. EFINUTRILES Study: Integrative Extra Virgin Olive Oil and Multimodal Lifestyle Interventions for Cardiovascular Health and SLE Management. Nutrients. 2025 Mar 19;17(6):1076. doi: 10.3390/nu17061076. PMID 40292522